CLINICAL TRIAL: NCT03021447
Title: Prediction of Postoperative Pain by Injection Pain of Propofol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, principal investigator, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-16-48
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative pain is a significant postoperative problem and it could be persistent if proper management is not provided. However, each patient shows different intensity of pain and different sensitivity to analgesics even if they underwent same procedures. Therefore, it would be useful to find the way to predict the postoperative pain sensitivity.

Propofol, a popular anesthetic agent, induces pain during injection, which can not completely prevented by opioid or lidocaine in some patients. This is considered to be related to patient's pain sensitivity and it might be associated with postoperative pain sensitivity.

Therefore, the relation of propofol injection pain and postoperative pain intensity will be explored.

ELIGIBILITY:
Inclusion Criteria:

* America Society of Anesthesiologists class I-II
* Laparoscopic cholecystectomy

Exclusion Criteria:

* Pregnancy
* Illiteracy

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for laparoscopic cholecystectomy will be included.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain intensity_1 | 10 min after postanesthesia care unit admission
  Postoperative pain will be evaluated with verbal numeric scale (0-10)

SECONDARY OUTCOMES:
postoperative pain intensity_2 | 20 min after postanesthesia care unit admission
  Postoperative pain will be evaluated with verbal numeric scale (0-10)
postoperative pain intensity_3 | 30 min after postanesthesia care unit admission
  Postoperative pain will be evaluated with verbal numeric scale (0-10)
postoperative pain intensity_4 | 4 hours after operation
  Postoperative pain will be evaluated with verbal numeric scale (0-10)
postoperative pain intensity_8 | 8 hours after operation
  Postoperative pain will be evaluated with verbal numeric scale (0-10)
postoperative pain intensity_12 | 12 hours after operation
  Postoperative pain will be evaluated with verbal numeric scale (0-10)
postoperative pain intensity_24 | 24 hours after operation
  Postoperative pain will be evaluated with verbal numeric scale (0-10)

IPD SHARING:
Plan to Share IPD: No